CLINICAL TRIAL: NCT05319860
Title: Effects of Aromatherapy on Chemotherapy-Induced Nausea and Vomiting: A Control Trial
Brief Title: Aromatherapy for Chemotherapy-induced Nausea and Vomiting (CINV)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Debbie Anglade, PhD, MSN, RN, Assistant Professor of Clinical, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20201412
Record Dates: First submitted 2022-03-31; First posted 2022-04-08 (Actual); Results first posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care With No Study Intervention (Active Comparator): Participants will receive standard medical care, consisting of antiemetic medicine at the first sign of Chemotherapy-Induced Nausea and Vomiting (CINV) on a schedule as prescribed by the healthcare provider.
  Interventions: Drug: Standard of Care Treatment for Chemotherapy Induced Nausea and Vomiting (CINV)
- Standard of Care With Study Intervention (Experimental): Participants will receive an aromatherapy inhaler for complementary in addition to their standard of care antiemetic medication for Chemotherapy-Induced Nausea and Vomiting (CINV).
  Interventions: Drug: Standard of Care Treatment for Chemotherapy Induced Nausea and Vomiting (CINV); Drug: Aromatherapy Care

INTERVENTIONS:
Drug: Standard of Care Treatment for Chemotherapy Induced Nausea and Vomiting (CINV) — Standard of care for CINV includes anti-nausea medication as needed after chemotherapy regimen given for up to 12 weeks.
Drug: Aromatherapy Care — An aromatherapy inhaler provided for use as needed after chemotherapy regimen given for up to 12 weeks. One normal inhale is equal to one dose of aromatherapy. Participants can use the aromatherapy as often as needed.
  Other Names: Soothing Scents QueaseEase aromatherapy inhalers
  Arms: Standard of Care With Study Intervention

SUMMARY:
The purpose of this study is to evaluate the use of aromatherapy to reduce nausea, vomiting, and the use of anti-emetic in cancer survivors undergoing moderate to highly emetogenic chemotherapy regimens.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Able to read and speak English or Spanish
3. Able to and willing to give informed consent
4. Currently undergoing moderate and high emetogenic chemotherapy (adjuvant or neoadjuvant)
5. Receiving three or more remaining cycles of chemotherapy
6. Symptoms of nausea or vomiting after the first chemotherapy infusion

Exclusion Criteria:

1. Unable or unwilling to give informed consent
2. Sensitivity to essential oils*
3. Olfactory disorders
4. Receiving chemotherapy for the first time
5. Undergoing low emetogenic chemotherapy regimens
6. Patients with hormone-sensitive cancers
7. Timely request of treating provider

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Debbie Anglade, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard of Care With No Study Intervention | Standard of Care With Study Intervention
Started | 48 | 52
Completed | 43 | 43
Not Completed | 5 | 9
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 3 | 1
Not completed — Withdrawal by Subject | 1 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care With No Study Intervention | Standard of Care With Study Intervention | Total
Number analyzed (Participants) | 48 | 52 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 39 | 44 | 83
  >=65 years | 9 | 8 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 35 | 60
  Male | 23 | 17 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 45 | 44 | 89
  Not Hispanic or Latino | 3 | 7 | 10
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 47 | 47 | 94
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Acute and Delayed Chemotherapy-Induced Nausea. The Self-reported Instruments Are Documented After the Chemotherapy Sessions and Collected on Study Visits 1, 2, and 3.
Description: Assessed by the mean/average score of the Multi Association of Supportive Care in Cancer (MASCC) Antiemesis tool (MAT). The scores were averaged across three visits to generate the reported values. The Antiemesis (MAT) tool is a user-friendly and reliable tool designed to measure acute and delayed Chemotherapy-Induced Nausea & Vomiting across patients' entire chemotherapy regimens. The acute phase is during the first 24 hours after receiving chemotherapy. The delayed phase is 2 to 4 days after chemotherapy treatment. The MAT tool assessment has a total score of 0-10 (how much nausea did you have over this period), with the higher scores indicating a higher level of nausea. The completed self-reported instruments were collected on study visits 1, 2, and 3, following their scheduled outpatient chemotherapy sessions. The participants' study visits 1, 2, and 3 schedules are based on their prescribed chemotherapy regimen duration, ranging from every two to four weeks for up to 12 weeks.
Time Frame: 24 hours and 2 to 4 days post chemotherapy on study visits 1, 2, and 3 every two to four weeks for up to 12 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard of Care With No Study Intervention | Standard of Care With Study Intervention
Number analyzed (Participants) | 48 | 51
score on a scale
  Acute Nausea (24 hours after chemotherapy begins) - MAT Question # 4 | 5.35 (0.30) | 4.57 (0.34)
  Delayed Nausea (4 days after chemotherapy begins)- MAT Question # 8 | 5.20 (0.30) | 4.55 (0.08)

2. Secondary Outcome: Change in Frequency of Antiemetic Medication Usage. The Self-reported Instruments Are Documented After the Chemotherapy Sessions and Collected on Study Visits 1, 2, and 3.
Description: Assessed by the average number of times antiemetic medications were used. The scores were averaged across three visits to generate the reported values. The completed self-reported instruments are collected on study visits 1, 2, and 3, following their scheduled outpatient chemotherapy sessions. The participants' study visits 1, 2, and 3 schedules are based on their prescribed chemotherapy regimen duration, ranging from every two to four weeks for up to 12 weeks.
Time Frame: Daily post-chemotherapy on study visits 1, 2, and 3 every two to four weeks for up to 12 weeks.
Measure: Mean (Standard Deviation); unit: average of medication use
Arm/Group | Standard of Care With No Study Intervention | Standard of Care With Study Intervention
Number analyzed (Participants) | 48 | 51
average of medication use | 9.89 (1.41) | 3.06 (0.35)

3. Primary Outcome: Acute and Delayed Chemotherapy-Induced Vomiting. The Self-reported Instruments Are Documented After the Chemotherapy Sessions and Collected on Study Visits 1, 2, and 3.
Description: Assessed by the mean/average score of the Multi Association of Supportive Care in Cancer (MASCC) Antiemesis tool (MAT). The MAT measures acute and delayed Chemotherapy-Induced vomiting (CINV) across patients' chemotherapy regimens using the question(s), "In the 24 hours since chemotherapy, did you have any vomiting?" and "Did you vomit 24 hours or more after chemotherapy?" respectively. Response options for both questions are a dichotomized Yes/No option. The percentage of participants who responded in the affirmative "Yes" were averaged with a score (ranging from 0-100%). The scores were averaged across three visits to generate the reported values. The completed self-reported instruments were collected on study visits 1, 2, and 3, following their scheduled outpatient chemotherapy sessions. The participants' study visits 1, 2, and 3 schedules are based on their prescribed chemotherapy regimen duration, ranging from every two to four weeks for up to 12 weeks.
Time Frame: 24 hours and 2 to 4 days post chemotherapy on study visits 1, 2, and 3 every two to four weeks for up to 12 weeks.
Measure: Mean (Standard Deviation); unit: percentage of participants
Arm/Group | Standard of Care With No Study Intervention | Standard of Care With Study Intervention
Number analyzed (Participants) | 48 | 51
percentage of participants
  Acute Vomiting-MAT | 11.1 (2.43) | 7.77 (3.95)
  Delayed Vomiting-MAT | 11.83 (4.79) | 5.95 (0)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Standard of Care With No Study Intervention | Standard of Care With Study Intervention
All-Cause Mortality (participants affected / at risk) | 1/48 | 1/52
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/52
Other Adverse Events (participants affected / at risk) | 0/48 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-13): https://cdn.clinicaltrials.gov/large-docs/60/NCT05319860/Prot_SAP_000.pdf